CLINICAL TRIAL: NCT05055323
Title: A Phase I Dose Escalation Study Using Pyrvinium Pamoate Targeting HuR in Pancreatic Ductal Adenocarcinoma
Brief Title: A Study to Determine if the Drug, Pyrvinium Pamoate, is Safe and Tolerable in Patients With Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20F.041; JT 14689 (Other: JeffTrial Number)
Record Dates: First submitted 2021-07-06; First posted 2021-09-24 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Resectable Pancreatic Ductal Adenocarcinoma; Stage 0 Pancreatic Cancer AJCC v8; Stage I Pancreatic Cancer AJCC v8; Stage IA Pancreatic Cancer AJCC v8; Stage IB Pancreatic Cancer AJCC v8; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pyrvinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pyrvinium pamoate) (Experimental): Patients receive pyrvinium pamoate PO QD for 3 days in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery.
  Interventions: Drug: Pyrvinium Pamoate

INTERVENTIONS:
Drug: Pyrvinium Pamoate — Given PO
  Other Names: 3546-41-6

SUMMARY:
This phase I trial studies the side effects and best dose of pyrvinium pamoate for the treatment of pancreatic ductal adenocarcinoma that cannot be removed by surgery (resectable). Pyrvinium pamoate may slow down tumor growth and help patients live longer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of pyrvinium pamoate (PP), dosed orally, in patients with pancreatic ductal adenocarcinoma (PDAC) that are surgical candidates.

SECONDARY OBJECTIVE:

I. Assessment of PP's pharmacokinetic and pharmacodynamic (PK/PD) profile and bioavailability in humans.

OUTLINE: This is a dose-escalation study.

Patients receive pyrvinium pamoate orally (PO) once daily (QD) for 3 days in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery.

After completion of study treatment, patients are followed up for 30 days and then every week for up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of pancreatic ductal adenocarcinoma (PDAC) suspected preoperatively who are deemed to be surgical candidates by the Thomas Jefferson University surgery department. Patients will be assessed by the pancreatic surgeons in the pancreatic surgery clinic, and if they are found to have resectable disease, they can be considered for this study
* Patients must not be on neoadjuvant therapy, or have received their last neoadjuvant treatment greater than or equal to within three weeks of starting PP therapy
* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Patients must have an estimated life expectancy of > 3 months, and Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* All patients regardless of age or gender must agree to observe proper contraceptive methods as to avoid becoming pregnant or causing pregnancy for the duration of the study (30 days after last dose of drug)

  * Males will practice safe sex methods (i.e. condoms)
  * Women of child bearing potential will practice safe sex methods (i.e. condoms, birth control), if a female on the study is of child-bearing age, they will have to take a urine human chorionic gonadotropin (HCG) (pregnancy) test prior to enrolling on the study

Exclusion Criteria:

* Patients with ongoing anticancer therapies, or those who will have received an anticancer therapeutic <3 weeks prior to the first dose of PP
* Any condition that precludes pancreatic surgical resection at the time of the study
* Pregnancy or currently breastfeeding
* Known allergic reactions to components of the study product(s): pyrvinium pamoate/ pyrvinium embonate (Molevac)
* Patients with chronic bowel conditions (such as inflammatory bowel disease (IBD))
* Kidney function impairment (serum creatine > 1.5 x ULN or creatine clearance </= 60 ml/1.73m^2 fr patients with creatine levels > 1.5 x ULN).
* Patients with liver function impairment: Alkaline phosphatase, ALT and AST above three folds the normal limit (see normal ranges); Total Bilirubin level > 3mg/dl; Albumin < 3g/dl

  * Alkaline phosphatase:
  * 0-9 years (yr): 83-280 IU/L at 37 degrees Celsius
  * 10-14 yr: 91-400
  * 15-17 yr: 37-240
  * 18-49 yr: 29-92
  * 50-74 yr: 25-120
  * 75-97 yr: 29-160
  * 98-99 yr: 29-120
  * > 99 yr: 29-160
* Patients with liver function impairment outside of the below ranges

  * Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]):

  ** Male (M): 1-45 IU/L at 37 degrees Celsius

  ** Female (F): 1-30
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]):

  * M: 7-42 IU/L at 37 degrees Celsius
  * F: 7-35
* Patients with liver function impairment outside of the below ranges

  * Albumin:
  * 0-1 yr: 2.6-4.4
  * 1-15 yr: 3.0-4.7
  * 16-99 yr: 3.2-4.9
* Patients with liver function impairment outside of the below ranges

  * Bilirubin, total:

  ** 0.1-0.9 mg/dL
* Patients with liver function impairment outside of the below ranges * Protein, total:

  * 0-1 yr: 4.6-7.2 g/dL
  * 1-15 yr: 5.7-8.2
  * 16-99 yr: 6.0-8.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limited toxicity (DLT) | Up to 30 days from last dose
  Considered any grade 3 or higher adverse event due to the drug itself or delay of surgery. Research coordinator will call patient every day to monitor for DLTs.

SECONDARY OUTCOMES:
Profile of pyrvinium pamoate (PP) | At Start of Treatment
  Will be assessed using liquid chromatography followed by mass spectrometry (LC/MS).
Profile of pyrvinium pamoate (PP) | Completion of treatment
  Will be assessed using liquid chromatography followed by mass spectrometry (LC/MS).
Bioavailability of PP | Up to 4 weeks
  Will be assessed using liquid chromatography followed by mass spectrometry (LC/MS).
Fatty tissue accumulation of PP | Up to 4 weeks
  Will be assessed using liquid chromatography followed by mass spectrometry (LC/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Harish Lavu, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ponzini FM, Schultz CW, Leiby BE, Cannaday S, Yeo T, Posey J, Bowne WB, Yeo C, Brody JR, Lavu H, Nevler A. Repurposing the FDA-approved anthelmintic pyrvinium pamoate for pancreatic cancer treatment: study protocol for a phase I clinical trial in early-stage pancreatic ductal adenocarcinoma. BMJ Open. 2023 Oct 17;13(10):e073839. doi: 10.1136/bmjopen-2023-073839. PMID 37848297